CLINICAL TRIAL: NCT00867763
Title: Clinical Research Study on in Vitro Maturation With IVF Compared to Mild Stimulation IVF
Brief Title: In Vitro Maturation With in Vitro Fertilization (IVF) Compared to Mild in Vitro Fertilization
Acronym: IVM vs IVF
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator changed location, requires new training effort
Sponsor: Batzofin Fertility Services (Other)
Responsible Party: Joe B. Massey MD, Massey
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2939
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2009-03

CONDITIONS: Infertility
Keywords: Polycystic ovaries,; Tubal occlusion; Unexplained infertility; Low ovarian reserve; Male factor infertility
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Fertilization in Vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVM (Experimental): Early egg retrieval, in vitro maturation, then IVF
  Interventions: Procedure: In vitro maturation and in vitro fertilization
- Mild IVF (Active Comparator): Mild gonadotropin and conventional IVF
  Interventions: Procedure: Low doses of gonadotropin stimulation.

INTERVENTIONS:
Procedure: In vitro maturation and in vitro fertilization — No gonadotropin, eggs harvested early
  Other Names: assisted reproduction
  Arms: IVM
Procedure: Low doses of gonadotropin stimulation. — Gonadotropin followed by conventional IVF
  Other Names: Assisted reproduction, IVF.
  Arms: Mild IVF

SUMMARY:
Methods of infertility treatment may involve in vitro fertilization or IVF. Though effective, IVF is complex and expensive. Methods using no gonadotropin hormone stimulation of the ovaries are being compared to mild stimulation doses. The goal of the research is to determine which of these if more suitable as a low cost approach for varying individual patients.

DETAILED DESCRIPTION:
Low cost environment is utilized, but fees are charged.

ELIGIBILITY:
Inclusion Criteria:

* Under age 42 female, normal uterine cavity, BMI 18-34kg/m2,

Exclusion Criteria:

* Donor eggs, donor sperm, myoma over 5 cm
* Current hydrosalpinx, abnormal uterine cavity.

Ages: 21 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1440 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Cost effectiveness | two years

SECONDARY OUTCOMES:
Ongoing pregnancy rates per cycle | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joe B Massey, MD, Principal Investigator — Batzofin Fertility Services
Locations (2):
- United States (2):
  - Batzofin Fertilty Services, New York, New York
  - BFS, New York, New York

REFERENCES:
- [Background] Son WY, Chung JT, Herrero B, Dean N, Demirtas E, Holzer H, Elizur S, Chian RC, Tan SL. Selection of the optimal day for oocyte retrieval based on the diameter of the dominant follicle in hCG-primed in vitro maturation cycles. Hum Reprod. 2008 Dec;23(12):2680-5. doi: 10.1093/humrep/den332. Epub 2008 Sep 4. PMID 18775885
- [Background] Son WY, Chung JT, Demirtas E, Holzer H, Sylvestre C, Buckett W, Chian RC, Tan SL. Comparison of in-vitro maturation cycles with and without in-vivo matured oocytes retrieved. Reprod Biomed Online. 2008 Jul;17(1):59-67. doi: 10.1016/s1472-6483(10)60294-5. PMID 18616892